CLINICAL TRIAL: NCT06494020
Title: Task Practice Combined With Transcutaneous Spinal Cord Stimulation to Reduce Muscle Co-contraction and Improve Motor Function in Chronic Spinal Cord Injury
Brief Title: Task Practice and Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: ONWARD Medical, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, James D. Guest, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20230228
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury Cervical; Spastic
Keywords: Transcutaneous; Transcutaneous Cervical Spinal Cord Stimulation
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Task Practice with stimulation (Experimental): Participants in this group will receive combined Transcutaneous cervical spinal cord stimulation with task practice for up to 2 months.
  Interventions: Other: Task Practice combined with Transcutaneous Spinal Cord Stimulation( TcSCS)

INTERVENTIONS:
Other: Task Practice combined with Transcutaneous Spinal Cord Stimulation( TcSCS) — Hand rehabilitative tasks ( for gross hand movement, grasp and pinch tasks) will be done by participants during which time the participant will receive TcSCS. This will be done three times a week for 60 minutes.

SUMMARY:
The goal of this study is to understand the effects of combined task practice with transcutaneous cervical spinal cord stimulation. The study will explore the effect of higher stimulation frequencies on spasticity. Transcutaneous stimulation has been shown to improve motor function in some individuals with chronic spinal cord injury. The study intends to explore scientifically the association between higher stimulation frequencies and spasticity/hypertonicity.

ELIGIBILITY:
Inclusion Criteria:

* 22-70 years of age
* Non-progressive cervical spinal cord injury
* Minimum 12 months year post-injury.
* American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification B, C, or D.
* Able to take part in upper extremity therapy procedures.
* GRASSP-Prehension score ≥10.
* MAS Score ≥3 but <6 in at least one arm.
* Can commit to the time required for the study.
* Stable medication profile for at least 4 weeks prior to enrollment.
* Able to reduce Baclofen dose to 30 mg or less daily.
* Capable of providing informed consent.

Exclusion Criteria:

* Has any unstable or significant medical condition that is likely to interfere with study procedures like severe neuropathic pain, depression, mood disorders, or other cognitive disorders.
* Has uncontrolled cardiopulmonary disease or cardiac symptoms.
* Requires ventilator support.
* Has been diagnosed with autonomic dysreflexia that is severe, unstable, and uncontrolled.
* Has an autoimmune etiology of spinal cord dysfunction/injury
* Previously diagnosed as having transverse myelitis
* History of additional neurologic diseases such as stroke, multiple sclerosis, traumatic brain injury, epilepsy or history of seizures.
* Peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.)
* Uncontrolled spasms, which have been unstable over the past three months prior to enrollment and are not expected to change.
* Received Botulinum toxin injections in their upper extremity, neck, or hand within six months prior to enrollment.
* Has painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or urinary tract infection at the time of enrollment.
* Breakdown in skin area that will come into contact with electrodes.
* Presence of syringomyelia as determined by an MRI.
* Currently undergoing treatment for cancer or has been in remission for less than 2 years.
* Received stem cell treatment within the past two years prior to enrollment.
* Has any active implanted medical device.
* Concurrent participation in another drug or device trial that may interfere with this study.
* In the opinion of the investigators, the study is not safe or appropriate for the participant.
* Persons who are unable to consent, pregnant women, and prisoners.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in motor performance as measured by The Graded Refined Assessment of Strength, Sensibility, and Prehension (GRASSP) test | baseline, up to 4 months
  GRASSP is a multimodal test that measures sensorimotor and prehension function in three domains that are important for the description of arm and hand functions, namely strength, sensation and prehension strength. It is an ordinal scale (minimum value = 0, maximum value = 100) with higher scores indicating better performance.
  There is a sensation category ordinal scale (minimum value = 0 maximum value = 24) that measures sensation where higher scores indicate greater sensation.
  The Prehension performance category has an ordinal scale (minimum value = 0 maximum value = 40) that measures prehension where higher scores indicate greater ability.

SECONDARY OUTCOMES:
Change in Spasticity as measured by Modified Ashworth Scale (MAS) | baseline, up to 4 months
  6 category ordinal scale (minimum value = 0 maximum value = 4) that measures spasticity where higher scores indicate greater spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: James Guest, MD, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami - Christine E. Lynn Rehabilitation Center, Miami, Florida
  - University of Miami, Miller School of Medicine, The Miami Project To Cure Paralysis, Miami, Florida

IPD SHARING:
Plan to Share IPD: No